CLINICAL TRIAL: NCT04394273
Title: The Effects of Exercise Training on Trunk Stabilizer Muscle Thickness, Functionality and Quality of Life During Pregnancy
Brief Title: The Effects of Exercise Training During Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Turkan Akbayrak, Professor, Hacettepe University
Other Study IDs: KA-19121
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Pregnancy
Keywords: pregnancy, exercise, stabilization
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 16 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Long- Term Exercise Group: They will exercise one an hour, two days a week, from the 16th week of pregnancy to the 32nd week (16 weeks).In this session, clinical pilates exercises are used as the basic exercise model and this exercise model is applied as a mixed exercise model in the form of posture and body mechanics training, lower-upper extremity strength training, pelvic floor muscle training and breathing exercises. Exercises can be started from the mat level and advanced in a modified manner with theraband and pilates ball.
  Interventions: Other: Exercise
- Short-Term Exercise Group: They will exercise half an hour, two days a week, from the 16th week of pregnancy to the 32nd week (16 weeks).n this session, clinical pilates exercises are used as the basic exercise model and this exercise model is applied as a mixed exercise model in the form of posture and body mechanics training, lower-upper extremity strength training, pelvic floor muscle training and breathing exercises. Exercises can be started from the mat level and advanced in a modified manner with theraband and pilates ball.
  Interventions: Other: Exercise
- Home Program: Pregnant women who choose the home program group are told to continue their home program until the 32nd week, which includes posture and body mechanics training, increase their physical activity levels and be as active as possible and take daily walks.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — stabilization exercise

SUMMARY:
Pregnancy is a physiological event that lasts for an average of 280 days or 40 weeks, starting with the embryo formed by the combination of ovum and sperm ready for fertilization. Many anatomical, physiological, social and psychological changes occur in the mother's body during pregnancy. In order to better adapt to these changes and to minimize problems during pregnancy, it is very beneficial for pregnants who do not have medical or obstetric risk to increase their physical activity level and exercise. Training programs created in light of the physical activity guidelines prepared specifically for the gestation period during pregnancy should be followed.

For this purpose, pregnant programs have been organized routinely as a group exercise two days a week in Hacettepe University, Physical Therapy and Rehabilitation Faculty, Women's & Men's Health Unit since 1990. The scope of this exercise program includes posture and body mechanics training, strengthening the lower and upper extremities, strengthening the abdominal and back muscles, pelvic floor exercises and breathing exercises. In one training session, 20 different exercises are performed and one session lasts about 60 minutes. For pregnant women with time limitations, sessions with less exercise and lasting about 30 minutes are held. Trainings are started in the 16th week of pregnancy and terminated in the 32nd week. Pregnant women who cannot participate in this group exercise program for personal reasons are given recommendations as home programs.

In the literature; There is no specific guide on the type of exercise, intensity, and frequency of the exercise that can affect the thickness of the trunk stabilizer muscles during pregnancy, improve functionality and quality of life. With this study, it is planned to investigate the effects of the exercise protocol applied on the thickness, functionality and quality of life of the body stabilizer muscles in pregnant women who routinely participate in the short or long group exercise program, which starts from the 16th week of pregnancy until the 32nd week of the week. In addition, the pregnant women, who could not participate in the short or long group exercise program and started their home program until the 32nd week of pregnancy and made their routine follow-ups, will be evaluated in the 16th and 32nd weeks of pregnancy.

At the end of this study; The change between body stabilizer muscle thickness, functionality and quality of life will be examined in three different groups, which continue routine short or long pregnant exercises and who can not participate in group exercise and follow up with the home program. In addition, data on trunk stabilizer muscle thickness, functionality and quality of life obtained from these three different groups will be compared. Thus, the literature will provide evidence of effective exercise protocols on trunk stabilizer muscle thickness, functionality and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Being in the 16th week of pregnancy
* Being literate
* Not having a history of abdominal surgeryExclusion Criteria:

Exclusion Criteri:

* Having one of the conditions such as heart disease, restrictive lung disease, cervical insufficiency, continuous bleeding in the second and third trimesters, placenta previa, risk of premature birth, membrane rupture, preeclampsia, and serious anemia.
* Not volunteering to participate in the study
* Not participating in more than 50% of long or short-term exercise sessions starting from the 16th week of pregnancy to the 32nd week (16 weeks) 2 days a week

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
thickness of trunk stabilizer muscles | 16-th week to 32-d week of pregnancy
  During the ultrasonography evaluation for the fetal development of the pregnant woman who came for routine obstetric examination, the pregnant women were lying in a supine position; Using 5-12 MHz linear probe (Logiq P5, General Electrics, Wisconsin, USA), rectus abdominis (at the level of umbilicus), transversus abdominis, external oblique and internal oblique (from the abdominal lateral) muscles will be bilaterally during axial imaging. Diaphragm thickness measurements will likewise be carried out through the mid-axillary line through the 7th intercostal space.
the degree of loss of functionality in low back pain | 16-th week to 32-d week of pregnancy
  Oswestry Disability Index will be used to evaluate the degree of loss of functionality in low back pain. Its validity and reliability in Turkish was determined in 2004 and consists of 10 items. The items question the severity of pain, self-care, lifting-carrying, walking, sitting, standing, sleep, the degree of pain change, travel and social life. When the total score is calculated, it is multiplied by two and said as a percentage. The maximum score is "100" and the minimum score is "0". As the total score increases, the level of disability increases.
The score of quality of life | 16-th week to 32-d week of pregnancy
  SF-36 will be used to determine the perceived quality of life in physical and mental health areas. SF-36 includes 36 questions and evaluation of eight health areas. These; physical functionality, physical role limitation, physical pain, general health, vitality, social functionality, emotional role restrictions and mental health. Scores from these subscales range from 0-100. "0" indicates poor health, "100" indicates goodness

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)